CLINICAL TRIAL: NCT06505395
Title: A Phase Ⅱ Randomized, Parallel-group, Open-label, Active-controlled Trial to Assess the Efficacy, Safety and Pharmacokinetics of the Long-acting Octreotide Subcutaneous Injection (SYHX2008) Versus Octreotide Microspheres (Sandostatin LAR@) in Patients With GEP-NET
Brief Title: A Trial to Assess Efficacy, Safety, Pharmacokinetics of Octreotide Subcutaneous Injection in Patients With Gastroentero-pancreatic Neuroendocrine Tumor (GEP-NET)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHX2008-004
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Neuroendocrine Pancreatic Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYHX2008 injection (Experimental)
  Interventions: Drug: SYHX2008 injection
- Octreotide Microspheres cohort (Sandostatin LAR@) (Active Comparator)
  Interventions: Drug: Sandostatin LAR@

INTERVENTIONS:
Drug: SYHX2008 injection — The patients will accept SYHX2008 injection by subcutaneous administration every cycle.
  Arms: SYHX2008 injection
Drug: Sandostatin LAR@ — The patients will accept Sandostatin LAR@ by intra-muscular administration every cycle.
  Arms: Octreotide Microspheres cohort (Sandostatin LAR@)

SUMMARY:
The purpose of this study is to compare the effectiveness, safety, pharmacokinetics (PK) of SYHX2008 vs Octreotide Microspheres (Sandostatin LAR@) in patients with advanced, well-differentiated GEP-NET.

DETAILED DESCRIPTION:
This is a Phase II, open-label randomized study to assess the PK, efficacy, and safety of SYHX2008 in adult patients with well-differentiated GEP-NET. Patients will be randomized to SYHX2008 cohort or Octreotide Microspheres cohort (Sandostatin LAR@).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years old;
2. Histologically confirmed, advanced GEP-NET;
3. At least 1 measurable, somatostatin receptor-positive lesion according to RECIST 1.1;
4. Previous treatment with ≤2 systemic antitumor drugs;
5. Patients who do not have liver metastasis, with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and alkaline phosphatase (ALP) levels ≤ 2.5 times the upper limit of normal (ULN) ; and who do have liver metastasis, with ALT and AST ≤ 5 times ULN; Serum total bilirubin <1.5 times the ULN; absolute neutrophil count (ANC) of ≥1.5×10^9/L, platelet count of ≥90×10^9/L, and hemoglobin ≥9 g/dL; or International Normalized Ratio (INR) ≤1.5 ULN and activated partial thromboplastin time (APTT) ≤1.5 ULN;
6. ECOG performance status of 0 to 1
7. Have expected survival of more than 3 months;
8. Adequately understand the study and voluntarily sign the Informed Consent Form;
9. Females patients with reproductive potential must agree to use an effective contraceptive method, for example, intrauterine devices, birth control medicine or condoms, during the study and within 3 months after study treatment discontinuation; or serum pregnancy tests negative and must be non-lactating participants; or males should agree contraception during the study and for within 3 months after study treatment discontinuation.

Exclusion Criteria:

1. Uncontrolled or severe diarrhea with significant dehydration;
2. Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection;
3. Anti-tumor therapy received within 4 weeks prior to the initiation of the investigational treatment, for example mammalian target of rapamycin (mTOR) inhibitors or multi-target tyrosine kinase inhibitors (TKI); or short-acting octreotide acetate was received subcutaneously or intravenously within 1 weeks prior to the initiation of the investigational treatment;
4. Interferon was received within 4 weeks prior to the initiation of the investigational treatment; or chemotherapy was received within 4 weeks prior to the initiation of the investigational treatment; or transarterial chemoembolization was received within 12 months prior to screening; or previously received peptide receptor radionuclide therapy (PRRT) at any time; or received radiation therapy, anti-tumor traditional Chinese medicine treatment, hepatic artery intervention embolization, liver metastasis cryoablation or radiofrequency ablation, and other systemic anti-tumor drug treatments within 4 weeks prior to the initiation of the investigational treatment; or had participated in other clinical trials within 30 days prior to screening
5. Surgery (except biopsy) within 28 days prior to the initiation of investigational treatment or unhealed surgical incision;
6. Glycated hemoglobin (HbA1c) > 8.5%;
7. Patients have symptomatic cholelithiasis or a history of symptomatic cholelithiasis at screening, but with no performed surgery treatment;
8. Patients with active brain metastases or cancerous meningitis meet any of the following criteria: a) Patients with prior brain metastases, imaging within 4 weeks prior to the first use of investigational drug show progression of the original lesion, or new brain metastases; b) Clinical symptoms associated with central nervous system metastasis did not recovery to baseline; c) Use cortisols, radiotherapy and other drugs to control the symptoms of central nervous system metastasis within 4 weeks before the first use of the investigational drug;
9. The adverse reactions of previous antitumor therapy have not returned to ≤ grade 1 according to CTCAE V5.0 (except that the investigators evaluate no safety risk, such as hair loss, grade 2 peripheral neuropathy or dysfunction);
10. Any clinically significant uncontrolled neurological, gastrointestinal, renal (serum creatinine > 1.5 ULN), pulmonary, or other significant disease requiring exclusion assessed in the opinion of the Investigator;
11. Patients had hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×10^4/ml or ≥2000 IU/ml); known Hepatitis C antibodies positive and HCV RNA higher than the lower detection limit ; or human immunodeficiency virus (HIV) positive, treponema pallidum antibody positive;.
12. A history of allergy to any excipient of the investigational drug or any similar chemical structure to the investigational drug;
13. Patients had any severe or uncontrolled disease, including: 1) poor blood pressure control (systolic ≥160 mmHg or diastolic ≥100 mmHg);2) grade I or higher myocardial ischemia or myocardial infarction, symptomatic or poorly controlled arrhythmia, or congenital long QT syndrome (including QTcF ≥450ms for males, QTcF ≥470ms for females), or ≥ Grade 2 congestive heart failure [NYHA classification]; 3) serious infections that are not under control (oral or intravenous systemic anti-infection therapy is required for 2 weeks before the first use of the investigational drug, except for uncomplicated urinary tract infections and upper respiratory tract infections);4) previous or current severe bleeding (>30ml of bleeding within 3 months), hemoptysis (>5ml of fresh blood within 4 weeks), or thromboembolic events (including transient ischemic attacks) within 12 months;
14. Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions are inappropriate for the use of the investigational product or affect interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as assessed by a Blinded Independent Review Committee (BIRC) | Up to 1 years following the last patient enrolled
  PFS is defined as time from the date of randomization to the date of the first documented disease progression as per RECIST 1.1 or death due to any cause (whichever occurs first)

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1 years following the last patient enrolled
  The time from the date of randomization to the date of death due to any cause
PFS as assessed by local Investigators | Up to 1 years following the last patient enrolled
  PFS as assessed by local Investigators
Overall response rate(ORR) | Up to 1 years following the last patient enrolled
  The proportion of patients with best overall response of complete response (CR) or partial response (PR), according to RECIST 1.1
Disease control rate (DCR) | Up to 1 years following the last patient enrolled
  The proportion of patients with a best overall response of CR, PR or stable disease (SD), according to RECIST 1.1
Duration of response (DOR) | Up to 1 years following the last patient enrolled
  The time from the date of the first documented response of CR or PR to the date of the first documented progression or death due to underlying cancer, according to RECIST 1.1
Time to Tomor Progression(TTP) | Up to 1 years following the last patient enrolled
  TTP is defined as time from the date of randomization to the date of the first documented disease progression as per RECIST 1.1
Control of cancer-like symptoms (diarrhea and/or flushing) | Up to 1 years following the last patient enrolled
  Assess the total occurrences of diarrhea and/or flushing ( cancer-like symptoms): Evaluate every 8 weeks (±3 days) for the first 12 months following the initial dosage, then every 12 weeks (±7 days). This assessment is based on the total instances of diarrhea and/or flushing episodes within the 7 days preceding the assessment visit.
Incidence of treatment-emergent adverse events | Up to 1 years following the last patient enrolled
  Incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, M.D, Study Chair — The First Medical Center, Chinese People's Liberation Army General Hospital, Beijing, China
Locations (1):
- Chinese PLA General Hosptial, Beijing, Beijing Municipality, China